CLINICAL TRIAL: NCT03129620
Title: Pharmacokinetics of Ampicillin in Neonates With Moderate to Severe Hypoxic-Ischemic Encephalopathy Undergoing Controlled Hypothermia
Brief Title: Pharmacokinetics of Ampicillin in Neonates With Moderate to Severe Hypoxic-Ischemic Encephalopathy
Status: Completed | Type: Observational
Sponsor: Drexel University (Other)
Responsible Party: Principal Investigator, Ogechukwu Menkiti, md, Drexel University
Other Study IDs: 1301001808
Record Dates: First submitted 2016-09-18; First posted 2017-04-26 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Hypothermia
Keywords: Ampicillin
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Controlled Hypothermia has become the standard of care for neonates with moderate to severe HIE. Ampicillin and aminoglycosides are drugs that are universally used for the treatment of suspected neonatal sepsis, which may or may not be responsible for the etiology of HIE. Currently, medication dosage regimens are not altered in the setting of CH. A better understanding of the effects of our interventions on this unique population may help us tailor our therapy to the specific circumstances of the patient

DETAILED DESCRIPTION:
Hypoxic-ischemic encephalopathy (HIE) affects approximately 1 to 2 per 1000 live births and remains a cause of significant morbidity and mortality in the neonatal period. In response to an anoxic insult, perfusion to vital organs is preserved; however, when this injury is profound concomitant injury to nonvital organs is observed. Controlled hypothermia (CH) has been accepted as a neuroprotective therapeutic modality for neonates with moderate to severe HIE because of its role in attenuating secondary brain injury. Neonates exhibit varying degrees of multiorgan dysfunction after a hypoxic-ischemic insult, although the added beneficial and potential adverse effects that CH has in these babies have not been completely delineated or understood.

CH has been shown to alter normal physiologic functioning of several organ systems. Specific physiologic changes as a consequence of CH have been demonstrated in both animal and human models. The observed reduction in cardiac output and reflexive increase in systemic vascular resistance in response to CH alter renal perfusion and subsequently reduce glomerular filtration . Drugs that are renally cleared may develop a prolonged half-life in this setting. Finally, drug metabolism may further be affected by altered hepatic blood flow and temperature-dependent effects on hepatic enzyme activity . Collectively, the potential effects of CH on drug metabolism and clearance are significant warranting further investigation. The investigator aims to evaluate the combined effects of hypoxia and hypothermia on ampicillin clearance and excretion

ELIGIBILITY:
Inclusion Criteria:

* Gestational age > 36 weeks
* Birth weight > 1800 grams
* Age < 6 hours old at the time of admission to the NICU
* Cord gas or ABG/VBG with pH < 7.0 or base deficit > 16 within the first hour of life
* Presence of seizures or evidence of moderate to severe encephalopathy
* Presence of central line for lab draws

Exclusion Criteria:

• Infants admitted for CH without central intravascular access.

Ages: 6 Hours to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates 0-24 hours of life
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2013-03; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Elevated ampicillin serum levels | 3 years
  Ampicillin concentration at 3 time points to determine clearance and serum levels

CONTACTS AND LOCATIONS:
Locations (1):
- St Christopher's Hospital for children, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No